CLINICAL TRIAL: NCT04918485
Title: Effect of Preoperative Psychological Intervention on the Degree of Cooperation During Tracheal Catheter Extubation in Patients Under General Anesthesia During Awakening Period
Brief Title: Effect of Preoperative Psychological Intervention on the Degree of Cooperation During Tracheal Catheter Extubation in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHZhejiangUChenshuyi
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-01

CONDITIONS: Nurse's Role

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group received psychological intervention (Experimental)
  Interventions: Other: preoperative psychological intervention
- the control group receive normal process before surgery (No Intervention)

INTERVENTIONS:
Other: preoperative psychological intervention — including closing the relationship between nurse and patient , knowledge education,
  Arms: the experimental group received psychological intervention

SUMMARY:
The patients in the experimental group received the relevant knowledge education in the recovery period 30 minutes before anesthesia. The operation time, anesthesia time, cooperation degree score, total cooperation rate and patient satisfaction were observed and recorded. Results: there was no significant difference in operation time and anesthesia time between the experimental group and the control group (P < 0.05). The percentage of patients in the experimental group was 20.12% and 70.89% respectively, while that in the control group was 40.32% and 20.73% respectively (P < 0.05). The total cooperation rate was 95.00% in the experimental group and 77.00% in the control group. There was significant difference between the two groups (P < 0.05). The satisfaction of patients in the experimental group was 95%. 65% of the patients in the control group were satisfied (P < 0.05). Conclusion: preoperative psychological intervention for patients with general anesthesia and endotracheal intubation can significantly reduce the restlessness and uncooperative phenomenon during extubation, and improve the cooperation rate and satisfaction of patients.

ELIGIBILITY:
Inclusion Criteria:

the patients who will undergo cholecystectomy surgery

Exclusion Criteria:

the patients who can not well communicate

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The total cooperation rate | through study completion, an average of half a year
  The total cooperation rate was 95.00% in the experimental group and 77.00% in the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd affiliated hospital, school of medicine, Zhejiang University, Hangzhou, Zhengjiang, China